CLINICAL TRIAL: NCT04870476
Title: "One Step at a Time" - an Internet-delivered Treatment for Patients Moderately Impaired by Bodily Distress Syndrome. A Feasibility Pilot Study
Brief Title: Feasibility and Acceptability of the Internet-delivered Treatment "One Step at the Time" for Bodily Distress Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: "During the feasibility study, it came to the research group's attention, that data was collected in an unauthorized manner. Therefore the trial has been terminated.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OneStep 1.0
Record Dates: First submitted 2020-02-17; First posted 2021-05-03 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Bodily Distress Disorder Moderate; Fibromyalgia; Chronic Fatigue Syndrome; Irritable Bowel Syndrome; Somatization Disorder
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Irritable Bowel Syndrome; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered treatment: "One step at the time" (Experimental): Internet-delivered treatment: "One step at the time". All participants receive the internet-delivered therapist-assisted 11-modules treatment program "One step at the time".
  Interventions: Behavioral: Internet-delivered treatment: "One step at the time"

INTERVENTIONS:
Behavioral: Internet-delivered treatment: "One step at the time" — The guided internet treatment program consists of 11 modules (+ 1 module for relatives) activated consecutively over a period of 14 weeks. The content is written psychoeducation, patient videos, audio exercises and exposure exercises. The program is therapist-guided; hence all patients will receive support primarily from a specific therapist during the 14 weeks.

SUMMARY:
This uncontrolled feasibility pilot study explores the acceptability and potential effect of a 14 week, 11-module, therapist-assisted, internet-delivered treatment program, "One step at the time", for patients moderately affected by Bodily Distress Syndrome. The study includes 25 participants aged 18-60 with multiple functional somatic symptoms for a duration of minimum 6 months. The focus of the feasibility trial is evaluation of treatment response, treatment satisfaction, program utility, recruitment and retention rates, data completion rates, and time requirement. The primary feasibility criterion is a +2.0 points change in patient-rated physical health measured by the SF-36 aggregate score physical health from before to after treatment.

DETAILED DESCRIPTION:
"One Step at the Time" - Internet-delivered Treatment for Patients Moderately Impaired by Bodily Distress Syndrome. A Feasibility Pilot Study.

Lisbeth Frostholm, Andreas Schröder, Johanne Liv Agger, Heidi Frølund Pedersen

Objective The objective of this uncontrolled pilot study is to test the feasibility of a future RCT by exploring the acceptability and effect of an internet-delivered treatment program, "One step at the time", for patients moderately affected by Bodily Distress Syndrome (BDS). The focus of the feasibility trial is evaluation of treatment response, treatment satisfaction, program utility, recruitment and retention rates, data completion rates, and time requirement. The primary feasibility criterion is an a priori defined change in patient-rated physical health from before to after treatment.

Design This study is designed as an uncontrolled, single-arm, single-center feasibility pilot study.

Participants The study includes 25 participants included from February to July 2020. The participants are recruited from The Research Clinic for Functional Disorders and Psychosomatics and The Pain and Headache Clinic, Aarhus University Hospital, Denmark, to which patients with multiple functional somatic symptoms are consecutively referred from GPs, medical specialists and hospital departments. Patients moderately affected by multiple symptoms are screened for eligibility by the eligibility criteria below. They undergo thorough diagnostic assessment by a medical doctor specialized in functional disorders after a thorough physical and psychological assessment including diagnostic interview (Schedules for Clinical Assessment in Neuropsychiatry), physical examination including blood pressure, blood test and a review of all medical records.

Eligibility criteria

Inclusion criteria:

1. Meet the diagnostic criteria for Bodily distress syndrome (BDS) with 2-3 of 4 symptom clusters
2. Moderate impact on daily life (self-reliant at home, can participate in activities outside the home)
3. Symptoms lasting for at least 6 months
4. 18-60 years at the time of inclusion

8. Previous stable educational or occupational attachment until at least 2 years prior to enrollment and expecting to return to occupational or educational activity 10. Motivation and time to participate in a psychological treatment program for treatment of BDS 11. IT skills and access to internet and computer/tablet 12. Willingness to engage in working with illness perception and behavioral change

Exclusion criteria:

5. Presence of other physical condition if the symptoms of this condition can not clearly be separated from symptoms of BDS or the condition is unstable/untreated 6. Current moderate or severe psychiatric disorder that substantially impacts daily life or demands special, individualized treatment, or clinical suspicion hereof, e.g. treatment-demanding depression or personality disorder 7. Current continuous treatment with opioids and drugs with opioid-like properties 9. Previous psychological treatment targeting BDS

Intervention "One step at the time" is a newly developed internet-delivered therapist-assisted treatment program for patients with BDS. The 11 modules + 1 module for relatives are primarily text-based but also contain audio files with guided exercises and videos with former patients. During a period of 14 weeks, patients are guided through the program modules assisted by a trained psychologist or psychiatrist.

Course If eligible and willing to participate, patients are included in the pilot study and assigned to a therapist (a trained psychologist or psychiatrist from The Research Clinic for Functional Disorders). Patients are contacted by telephone by the therapist and guided to login to the program platform and initiate treatment. The therapist follows the patient through the 11 treatment modules and provides guidance when needed. Patients and therapists primarily communicate through asynchronously written messages, and occasionally by telephone. Treatment duration is 14 weeks.

Measurements Patient-rated outcome measures are collected through a web-based program at the time of screening (before inclusion) (T0, baseline), before treatment (T1, 2 weeks), at end of treatment (T3, 16 weeks) and at 3 months after treatment (follow-up, 28 months) (T4). Clinician-rated outcome measures are collected at the time of diagnostic assessment and at end of treatment.

Patient-rated measures include:

* physical, mental, and social health measured by SF-36 with emphasis on the aggregate score physical health
* overall health improvement measured by the 5-point clinical global improvement scale (CGI)
* symptom intensity and symptom interference measured by The Numeric Rating Scale
* symptoms of anxiety, depression, and somatization measured by relevant subscores of the 92-item Danish version of the Symptom Checklist (SCL-92)
* bodily symptoms measured by The BDS Checklist
* illness worry measured by Whiteley-7
* illness perception measured by Brief-IPQ
* illness behaviour measured by BRIQ
* sense of meaningfulness measured by The Sources of Meaning and Meaning in Life Questionnaire (SoMe short version)
* treatment expectancy, rationale credibility, and treatment satisfaction measured by the credibility/expectancy questionnaire
* work performance and work absence measured questionnaire for Costs associated with Psychiatric Illness (TiC-P)
* demographic variables
* negative effects of psychotherapy measured by the inventory for the assessment of negative effects of psychotherapy (INEP)
* program utility measured by the Internet Evaluation and Utility Questionnaire
* patients' experience and satisfaction with assessment and treatment measured by questionnaires and qualitative semi-structured interviews

Other measures include:

* clinician-rated improvement measured by the 5-point clinical global improvement scale (CGI),
* therapist time spent per patient
* clinician-rated program utility measured by the Internet Evaluation and Utility Questionnaire
* recruitment and retention rates and data completeness.

Feasibility outcomes

1) Changes in patient-rated physical health from before to after the treatment measured by the SF-36 aggregate score Physical Health.

1. Recruitment and retention rates, time requirements and data completeness as measured by the rate of eligible patients willing to participate, the rate of included patients completing the treatment program (defined as completion of at least 5 modules), therapists' time spent per patient, and the rate of treatment completers providing full data.
2. Patients' treatment satisfaction and assessment of program utility as measured by the credibility/expectancy questionnaire, a patient satisfaction questionnaire and the internet evaluation and utility questionnaire.
3. Patients' and therapists' impression of treatment effect as measured by the clinical global improvement 5-point Likert scale).

Feasibility criteria

We regard a future study testing the treatment program "One step at the time" in an RCT as feasible if:

1. A mean change in the SF-36 aggregate score Physical Health is at least +2.0 points from baseline (T0, baseline) or inclusion (T1, 2 weeks) to end of treatment (T2, 16 weeks) for treatment completers.
2. 75% of the patients included in the study complete the treatment program (defined as completion of at least 5 of 11 modules) and 90% of treatment completers provide full data

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for Bodily distress syndrome (BDS) with 2-3 of 4 symptom clusters
2. Moderate impact on daily life (self-reliant at home, can participate in activities outside the home)
3. Symptoms lasting for at least 6 months
4. 18-60 years at the time of inclusion
5. Previous stable educational or occupational attachment until at least 2 years prior to enrollment and expecting to return to occupational or educational activity
6. Motivation and time to participate in a psychological treatment program for treatment of BDS
7. IT skills and access to internet and computer/tablet
8. Willingness to engage in working with illness perception and behavioral change

Exclusion Criteria:

1. Presence of other physical condition if the symptoms of this condition can not clearly be separated from symptoms of BDS or the condition is unstable/untreated
2. Current moderate or severe psychiatric disorder that substantially impacts daily life or demands special, individualized treatment, or clinical suspicion hereof, e.g. treatment-demanding depression or personality disorder
3. Current continuous treatment with opioids and drugs with opioid-like properties
4. Previous psychological treatment targeting BDS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in physical Health | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 months)
  Patient-rated physical health measured by the SF-36 aggregate score Physical Health

SECONDARY OUTCOMES:
SF-36 physical health | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Changes in physical, mental, and social health
5-point clinical global improvement scale (CGI) | after treatment (14 weeks)
  Overall health improvement
The Numeric Rating Scale | every 2 weeks during treatment
  Changes in symptom intensity and symptom interference
Relevant subscores of the 92-item Danish version of the Symptom Checklist (SCL-92) | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Changes in symptoms of anxiety, depression, and somatization
The BDS Checklist | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Symptom checklist
Whiteley-7 | Baseline, before treatment, after treatment and at 3 month follow up
  Changes in illness worry
Brief-Illness perception questionnaire | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Changes in illness perception
The Behavioural Responses to Illness Questionnaire (BRIQ) Changes in illness behaviour | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Changes in illness behaviour
The credibility/expectancy questionnaire | Before treatment (2 weeks) and after treatment (16 weeks)
  Treatment expectancy, rationale credibility, and treatment satisfaction
Costs associated with Psychiatric Illness (TiC-P) | Before treatment (2 weeks) and at 3 month follow up (16 weeks)
  Changes in work performance and work absence
The inventory for the assessment of negative effects of psychotherapy (INEP) | After treatment (16 weeks)
  Negative effects of psychotherapy
The Internet Evaluation and Utility Questionnaire | after treatment (16 weeks)
  Program utility
The Sources of Meaning and Meaning in Life Questionnaire (SoMe short version) | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Chnages in sense of meaningfulness and crisis of meaning

OTHER OUTCOMES:
Patients' experience and satisfaction with assessment and treatment | During treatment
  Qualitative semi-structured interviews
5-point clinical global improvement scale (CGI) | After treatment (16 weeks)
  Clinician-rated improvement
Therapist time spent per patient | During treatment
  Time spent per patient
The Internet Evaluation and Utility Questionnaire | After treatment (16 weeks)
  Clinician-rated program utility
Recruitment and retention rates and data completeness. | Baseline, before treatment (2 weeks), after treatment (16 weeks) and at 3 month follow up (28 weeks)
  Rates of eligible patients willing to participate, completion rate (at least 5 modules) and data completeness.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Frostholm, PhD, Principal Investigator — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: No